CLINICAL TRIAL: NCT00618904
Title: Clinical Efficacy of Probiotic Bacteria in Subjects With Irritable Bowel Syndrome (IBS), Functional Diarrhea, or Functional Bloating
Brief Title: Efficacy of Probiotic Bacteria in Subjects With IBS or Functional Diarrhea/ Bloating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Danisco (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 04-1704
Record Dates: First submitted 2008-02-07; First posted 2008-02-20 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-07

CONDITIONS: Pain
Keywords: Probiotics; Functional Gastrointestinal Symptoms
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Probiotic containing Lactobacillus and Bifidobacterium
  Interventions: Dietary Supplement: Probiotics - Lactobacillus and bifidobacterium
- 2 (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics - Lactobacillus and bifidobacterium — Probiotics administered bid for 6 weeks.
  Arms: 1
Dietary Supplement: Placebo — Placebo administered bid for 6 weeks.
  Arms: 2

SUMMARY:
To determine if probiotics bacteria, specifically lactobacillus and bifidobacterium, improve gastrointestinal symptoms in patients with IBS, functional diarrhea, or functional bloating.

DETAILED DESCRIPTION:
Functional Bowel disorders (FBD) including Irritable Bowel Syndrome (IBS) are characterized by a variable combination of chronic or recurrent gastrointestinal symptoms not explained by structural or biochemical abnormalities. IBS is the most common functional gastrointestinal disorder, affecting 8% to 23% of adults in the western world and accounts for 12% of primary care and 28% of gastroenterological practice visits yearly. The pathophysiology of IBS is not completely understood and currently available drug treatments for IBS are very limited (1-2). The apparent success of the use of probiotics in several gut disorders (e.g., IBD) together with the greater understanding of the role of inflammation and intestinal microflora in the pathophysiology of IBS has led to increased interest in use of probiotics in patients with IBS (3). The data on the use of probiotic in IBS is limited. However, few reported studies show encouraging results and suggests some symptomatic response and parallel improvement in quality of life (3-4). A controlled, double-blind study, randomized 20 patients with IBS to L. plantarum 299v or placebo for 4 weeks concluded that L. plantarum decreased abdominal pain and tended to normalize stool frequency in constipated patients (5). On the other hand, Lactobacillus casei GG, was found to improve stool consistency in patients with IBS and diarrhea (6). A recent randomized controlled trial using the probiotic formulation VSL#3 improved abdominal bloating in patients with diarrhea-predominant IBS. However, no differences in gastrointestinal transit measurement, bowel function scores or satisfactory global symptom relief were shown (7). The inconsistent findings of these clinical studies may be accounted to the differences in probiotics composition and the heterogeneous and multifactorial nature of the disorder. However, these studies indicate a potential relationship between probiotics therapy and functional abdominal symptoms and suggesting that the possible role of probiotics in the treatment of IBS deserves further study.

ELIGIBILITY:
Inclusion Criteria:

* The subject is 18 to 75 years old.
* The subject is an ambulatory outpatient.
* The subject has IBS, or functional diarrhea, or functional bloating according to the Rome II criteria for functional GI disorders.
* The subject has the above symptoms for at least two weeks, despite current therapy. For diarrhea, we will use the definition of a mean of >2 bowel movements per day, or a mean score of > 4 on the Bristol Stool Form Scale per week. For bloating we will use the Rome II definition "a feeling of abdominal fullness or bloating".
* Subject must have had a colonoscopy if age > 50y/o.
* The subject's symptoms are mild to moderate symptoms in severity. Symptoms severity will be assessed at baseline and at the end of the 2-weeks screening period to determine eligibility prior randomization. Severity of bowel symptoms will be determined using the Francis Whorwell IBS severity scale: Mild <175, Moderate 175-300, Severe >300

Exclusion Criteria:

* The subject has inflammation or structural abnormality of the digestive tract (e.g. inflammatory bowel disease (IBD), duodenal ulcer (DU) or gastric ulcer (GU), obstruction, symptomatic cholelithiasis).
* The subject has severe FBD related symptoms at baseline.
* The subject has a serious, unstable medical condition.
* The subject has insulin-dependent Diabetes Mellitus.
* The subject had a major psychiatric diagnosis or a suicide attempt within the last two years.
* The subject has a history of alcohol or substance abuse within two years.
* The subject has abnormal laboratory results (including ALT or AST > than 2.5 times normal, serum creatinine >2.0mg/dl, untreated abnormal TSH value)
* The subject has been treated for a malignancy within the last 5 years (except BCC or SCC skin cancer).
* The subject has been diagnosed with lactase deficiency and this can explain their symptoms (i.e., symptoms resolved or reduced significantly with lactose-free diet.)
* The subject has participated in a drug study within the last 21 days.
* The subject received antibiotic treatment during the last 8 weeks. (If the subject was on antibiotic treatment, a washout period of 8 weeks is required).
* The subject had previous significant intestinal surgery.
* The subject is pregnant or lactating, or unwilling to maintain effective contraception during course of study
* The subject is predisposed to infection (i.e. their immune system is compromised, they have rheumatic heart disease, an artificial valve, history of bacterial endocarditis, or an active bacterial disease)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2005-12; Primary Completion 2007-02 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be the global relief of GI symptoms as assessed by Global Symptom Assessment (GSA) of relief of functional GI symptoms.

SECONDARY OUTCOMES:
Assess the improvement of specific functional bowel disorders (FBD) related symptoms and Health Related Quality of Life (HRQOL).

CONTACTS AND LOCATIONS:
Overall Officials: Yehuda Ringel, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Ringel-Kulka T, Palsson OS, Maier D, Carroll I, Galanko JA, Leyer G, Ringel Y. Probiotic bacteria Lactobacillus acidophilus NCFM and Bifidobacterium lactis Bi-07 versus placebo for the symptoms of bloating in patients with functional bowel disorders: a double-blind study. J Clin Gastroenterol. 2011 Jul;45(6):518-25. doi: 10.1097/MCG.0b013e31820ca4d6. PMID 21436726